CLINICAL TRIAL: NCT04695145
Title: A Randomized Pilot Study Comparing Vigorous Group Aerobic Exercise vs. Group Leisure Activities for Mild to Moderate Depression in Adolescents
Brief Title: Aerobic Group Exercise for Adolescents With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Region Halland (Other); Halmstad University (Other); The Rydberg Laboratory for Applied Sciences, Halmstad, Sweden (Unknown); Karolinska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-03364
Record Dates: First submitted 2020-12-02; First posted 2021-01-05 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Depressive Disorder, Major
Keywords: adolescent; depression; exercise intervention; biomarker; cost evaluation; qualitative
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Exercise; Population Groups

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study - pilot version
Who Masked: Outcomes Assessor
Masking Description: The baseline and outcome assessor is not working at the clinic and is not informed of treatment mode. The patient is informed at the beginning of the interview not to disclose any information about mode of treatment. All interviews are recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise in group (Experimental): The patients will participate in aerobic group exercise for 60 minutes three times a week for 12 weeks with continuous heart rate monitoring. The sessions will be held in a small gym under supervision of a personal trainer with special training in medical issues. The exercise will be monitored with continuous heart rate registration.
  The group training session will begin with a warm-up to increase heart rate including balance tasks and dynamic stretching for 10-15 minutes. Every third session will be pure aerobic training, every third session will be strengthening exercises designed to also increase heart rate, and every third session will be a mixed session of both aerobic and strength exercises. All major muscle groups will be used at each session. Interval training with gradually increased intensity throughout the program will be applied.
  Interventions: Behavioral: Aerobic exercise in group
- Group sessions with leisure activities (Active Comparator): The control group will receive leisure activity in a group setting for one hour three times a week for 12 weeks. The sessions will be held at the same weekdays and about the same hours as the exercise group sessions. The same group leaders as in the exercise sessions will participate in leisure sessions and will support the adolescents through reminders and reassurance before and during the sessions to enhance adherence. The sessions will start with a check in on feelings, recent events and difficulties (i.e. supportive listening but not any interventions) followed by non heart rate increasing activities, such as playing games or watching movies together.
  Interventions: Behavioral: Group sessions with leisure activities

INTERVENTIONS:
Behavioral: Aerobic exercise in group — Progression
  The goal with every new week should be making every workout a little bit harder than the week before.
  Strength sessions
  * Week 1-6: 12-18 reps x 2 set per exercise and muscle 30 s rest between exercises
  * Week 7-12: 10-12 reps x 3 set per exercise and muscle 20 s rest between exercises
  Adding weight with gym equipment or changing body position in the exercises to succeed with the rep scheme and making it harder as the group develop their physical and mental ability.
  Conditioning sessions
  * Week 1-6: 75 seconds work time x 1 set per exercise 30 seconds of rest between exercises
  * Week 7-12: 50 seconds work time x 2 set per exercise 20 seconds of rest between exercises
  Mixed sessions
  * Week 1-6: 35 s work time per exercise 25 s rest between exercises x 2 rounds
  * Week 7-12: 45 s work time per exercise 15 s rest between exercises x 2 rounds
  Arms: Aerobic exercise in group
Behavioral: Group sessions with leisure activities — The control group will receive leisure activity in a group setting for one hour three times a week for 12 weeks. The sessions will be held at the same weekdays and about the same hours as the exercise group sessions. The same group leaders as in the exercise sessions will participate in leisure sessions and will support the adolescents through reminders and reassurance before and during the sessions to enhance adherence. The sessions will start with a check in on feelings, recent events and difficulties (i.e. supportive listening but not any interventions) followed by non heart rate increasing activities, such as playing games or watching movies together.
  Arms: Group sessions with leisure activities

SUMMARY:
The aim is to evaluate aerobic group exercise versus leisure group activities in adolescents with mild to moderate depression.

Primary outcome is Children's Depression Rating Scale - Revised (CDRS-R). Secondary outcomes are Clinical Global Impressions - Severity and Improvement scales (CGI), self-reported Quick Inventory of Depression Symptomatology (QIDS- A17-SR), the self-reported Outcome Rating Scale (ORS), clinician rated Children Global Assessment Scale (C-GAS), aerobic capacity (VO2max), muscular strength, body, Body Mass Index (BMI), presence or activity of selected biological markers of neuroprotection and neuroinflammation in blood samples and a cost evaluation rated by parents with Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness - Child version (Tic-P). Further objectives are qualitative interviews to explore adolescents' experiences of the intervention as well as how their health and lifestyle are influenced and a validation of QIDS- A17-C and QIDS- A17-SR versus CDRS-R will be performed.

DETAILED DESCRIPTION:
Detailed Description: Depression is common in adolescence and prevalence is increasing. It is a major cause of disability in adolescents worldwide and contributes to lower educational achievements, increased risks of substance abuse, suicide and a risk factor for cardiovascular disease. The effect of evidence based treatments with antidepressants or psychotherapy such as cognitive behavioural therapy (CBT) or interpersonal therapy (IPT) are modest. Selective serotonin uptake inhibitors (SSRIs) have shown effect on depression in children and adolescents, but the effect is often insufficient.

Aerobic exercise seems to have effect on depression in adolescents but studies have several shortcomings. Recruitment was mostly in non-clinical or primary care facilities, results are heterogeneous and adequate control groups are lacking. More data on qualitative, cost-effectiveness and biomarker aspects are clearly warranted.

Objectives

1. Primary objective To evaluate aerobic group exercise versus leisure group activities on clinician rated depression symptoms among adolescents in child and adolescent outpatient care with mild to moderate depressive disorder by measuring changes in Children's Depression Rating Scale- Revised (CDRS-R).
2. Secondary objectives Secondary objectives are clinician rated Clinicial Global Impression - Severity (CGI-S) and Improvement scales (CGI-I) and function with Children Global Assessment Scale (C-GAS), self-rated symptoms (QIDS-A17-SR) and function with the Outcome Rating Scale (ORS), aerobic capacity measured by a submaximal aerobic capacity test, muscular strength measured by the isometric mid-thigh pull strength test, a hand grip strength test and muscular endurance by the one-leg sit-to-stand test, and body composition with a bioelectrical impedance analysis and presence or activity of selected biological markers of neuroprotection and neuroinflammation in blood samples.

Moreover, the investigators will assess cost-effectiveness in this trial. Another secondary objective is to explore adolescents' experiences of the intervention as well as how their health and lifestyle are influenced by the intervention through qualitative interviews. Finally, we will validate the QIDS- A17-C and QIDS-A17-SR against CDRS-R.

The statistical power of this trial is not designed to arrive at significant findings, but to validate the measures and data collection approach and to gather preliminary data to inform the power analysis when planning the full-scale RCT.

Project description

1. Design The study will be a one-sited randomized pilot study that will include 24 adolescents with ongoing mild to moderate depression after three or more visits and brief psychosocial interventions. Participants will be randomized to receive 12 weeks of either aerobic group exercise or leisure group activities at a ratio of 1:1. Adolescents allocated to leisure activities will get the opportunity to participate in aerobic exercise after the evaluation at 13 weeks and at a one-year follow up.
2. Control group justification By using leisure activities in a group setting as a control group, the investigators control for the possible effect on social interaction and behavioural activation.
3. Study setting The study will be conducted at the child and adolescent psychiatric clinic in Halmstad. The site is the only provider of specialised care for adolescent depression in a small city with surrounding countryside with about 7500 adolescents. Outcome variables are assessed by communicating with patients on smart phones. Research interviews will be recorded video calls, and self-rated measures will be collected electronically.
4. Power analysis Not applicable in a pilot trial
5. Data collection QIDS-A17-SR and K-SADS-PL with the adolescent and parent will be conducted at the clinic before baseline. CDRS-R, QIDS-A17-C and CGAS at baseline, 13 weeks, 26 weeks (for controls that exercise after the initial 12 weeks) and one- year follow up assessment will be conducted through a recorded video call. Patients fill out a web based questionnaire with QIDS-A17-SR and ORS every two weeks during the 12 weeks intervention period and monthly during the follow-up until one year.
6. Screening and recruitment procedures The investigators will recruit patients from child and adolescent psychiatric outpatient care in Halmstad diagnosed with depression and who have had at least three visits and thus most likely have received some basic psychosocial interventions. The patients will be identified through a scanning of the outpatient computer system or identified by staff.
7. Randomisation, enrolment and masking. Participants will be randomized at a ratio of 1:1 to aerobic group exercise or group leisure activities. Sealed envelopes with randomisation numbers will be stored in a locked cabinet. Randomization will occur in slots of 8 patients to give equally sized groups if full inclusion is not possible within the set time frame.

   The investigator (TC) conducting the baseline and 13 week evaluation will be blind to treatment allocation. The outcome measures are identical for the two groups, ensuring that the assessors remain blind. Participants will be reminded at the start of each interview not to reveal their arm of allocation. To measure blinding integrity, the assessor will record whether the participating families inadvertently reveal their group allocation. At the one-year open follow up, all patients have had the opportunity to exercise and the evaluation is unblinded.
8. Rater training Research TC will get instructions and perform CDRS-R supported by an experienced user of CDRS-R including rating and discuss four recorded videos.
9. Baseline assessments Clinician video evaluation: CDRS-R, QIDS-A17-C, CGI and C-GAS CDRS-R, QIDS-A17-C and C-GAS will be conducted through a recorded video call. Inter rater test will be performed between RW, TC and PI on ten CDRS-R, C-GAS and QIDS-A17-C from baseline.

   * Self-reported web based: QIDS-A17-SR and ORS
   * Parent cost evaluation with Tic-P
   * Measures at site: aerobic capacity, muscular strength and body composition.
   * Blood sampling
10. Recurrent evaluation. QIDS-A17-SR and ORS will web-based be filled in every other week. After two weeks of intervention also questions on safety, side effects and treatment credibility.
11. 13 week evaluation

    * Clinician video evaluation: CDRS-R, CGI and C-GAS
    * Self-reported web based by ES-maker: QIDS-A17-SR and ORS
    * Parent rated and web-based cost evaluation with Tic-P
    * Qualitative interviews with participants according to interview guide
    * Anthropometric measures at site: height, weight, aerobic capacity, muscular strength and body composition.
    * Blood sampling
12. End of trial. The trial will end when the final data from the one-year follow up has been collected for the last patient.
13. Participant withdrawal. Participants are free to withdraw from the trial at any point. After the withdrawal, participants will not be requested to complete any further measures, but will be asked to provide non-obligatory feedback regarding their reason for withdrawal Once participants have withdrawn from the trial, it will not be possible to re-enter or resume treatment. Withdrawn patients will not be replaced in the trial.
14. Concomitant interventions. Medication for depression is required to have been stable four weeks prior to inclusion. Medications with stimulants or neuroleptics need to have been stable for two weeks. Additionally, the participants are encouraged not to alter his/hers medication or receive any psychological treatment until after the 13 week evaluation. Visits for safety evaluations, for school-planning and to issue parental child-sick leave are permitted.
15. Data management. All aspects of data management of the trial will comply with the General Data Protection Regulation (GDPR). Notes will be made in the clinical records.
16. Statistical analyses. Statistical Package for the Social Sciences (SPSS) version 24 will be used for analyses. Multilevel regression modelling will be performed to quantify the treatment effects on the change scores from baseline measures with included explanatory variables.
17. Adverse events.

    Serious Adverse Event (SAE) is any unfortunate occurrence that:
    * results in death
    * is life-threatening
    * requires hospitalisation
    * results in persistent or significant disability or incapacity
    * is otherwise considered medically significant by the investigator

    Suspected Unexpected Serious Adverse Reaction (SUSAR) is any SAE that is deemed to be:
    * related to the trial intervention AND
    * unexpected AND
    * Not listed in the protocol as an expected adverse event of the intervention Expected adverse events

    The investigators have considered the following events as possible adverse events:
    * Increased depressive symptoms
    * Suicide attempt
    * Increased stress due to time consuming sessions and transportation
    * Injuries due to exercise The investigators also have to consider that psychological adverse events may also be symptoms of the underlying condition, i.e. depressive disorder, rather than the intervention itself.

    The assessment of the relationship between adverse events and the administration of the treatment is a decision based on all available information. The final decision is taken by the PI. If the event is a result of the administration of any of the research procedures then it will be classified as related.

    If the event has been listed in the protocol as an expected side effect of the intervention then the event will be classified as expected. If the event is not listed then it will be classified as unexpected.

    All adverse events will be noted by the trial coordinator in a specific log (including date, recorded clinical symptoms, and a brief description of the event). SAEs and SUSARs will be recorded in the trial coordinator's log. Appropriate action will be taken in the case of SAE and SUSAR, making sure the participant will get in contact with suitable health care services. Events will be considered as potentially treatment-related up to the 13 weeks evaluation and for the control group up to 26 weeks, where the reporting of adverse events will terminate.
18. Notification of serious breaches to GCP and/or the protocol

    A "serious breach" is defined as a breach which is likely to a significant degree affect:
    * the safety or physical or mental integrity of participants or
    * the scientific value of the trial. The PI will notify the Ethical Review Board in writing of any serious breach. Reports of serious breaches will contain when the breach occurred, the location, who was involved, the outcome and any information given to participants. An explanation regarding the cause of the serious breach will be given, and the Ethical Review Board will be informed of planned further actions.
19. Data sharing The investigators will not share trial data with other researchers around the world.
20. Ethical considerations The study has been approved by the National Ethical Review Board in Sweden. All patients and parents will be provided by oral and written information about the study. Informed consent in writing will be provided from patients and parents to participants below 15 years of age.

    Participants randomised to leisure activities will get the opportunity to exercise after 13 weeks, ensuring all participants are offered the active treatment.
21. Implications Aerobic group exercise can, if shown to be effective, become a recommended treatment option for major depressive disorder in adolescents either alone or as an addition to present treatment options with cognitive behavioural therapy and antidepressants.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 mild to moderate depression
* Who have received evaluation and basic psychosocial interventions for 4-8 weeks (minimum four visits) without response, i.e. not achieved improvement by at least 50 % as assessed from clinical records

Exclusion Criteria:

* Eating disorder
* High risk for suicide
* Intellectual disability
* Actual physical activity the last four weeks meeting the level for sustained health by American College of Sports Medicine, i.e. at least 150 min per week of moderate intensity or 75 min per week of high intensity38
* Adjustment of antidepressant medication within the last four weeks or stimulants the last two weeks
* Chronic somatic illness precluding exercise
* In need of interpreter
* Social circumstances interfering with a regular exercise schedule
* Concomitant psychotherapy

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Children's Depression Rating Scale- Revised (CDRS-R) | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Clinician administered interview about symptoms of depression, range 17 (best) - 113 (worst)

SECONDARY OUTCOMES:
Change in Quick Inventory of Depressive Symptomatology-Self Rated (QIDS-A17-SR) | Every two weeks during the 12 week intervention and monthly during the preceding year.
  Self report form about symptoms of depression, range 0 (best) - 27 (worst)
Change in Children Global Assessment Scale (C-GAS), | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Clinician administered interview about psychosocial function, 1(worst) - 100 (best)
Change in Outcome Rating Scale (ORS) | Every two weeks during the 12 week intervention and monthly during the preceding year.
  Self report form about psychosocial function, range 1 (worst) - 100 (best)
Change in Aerobic capacity | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Submaximal and maximal aerobic capacity test, measured as Oxygen consumption (ml) / weight (kg) x time (minute), range typically about 20 (lowest) - about 60 (highest)
Change in Muscular strength | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Change in Isometric mid-thigh pull strength test (kg), a hand grip strength test (kg) and muscular endurance by the time to repeat 5 one-leg sit-to-stand test (seconds), and body composition with a bioelectrical impedance analysis (resistance in Ohm, lower value indicates increase in muscle and higher value increase in fat)
Change in Biological markers of neuroprotection and neuroinflammation in blood samples | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Biomarkers for neuroprotection (higher value is better) and neuroinflammation (lower value is better) will be analysed: BDNF, CRP, IL-6, KYNA/3HK75, KYNA/QUIN75, KYN-ACID75, SIL-2 receptor, TNF-alpha, IGF-1 and their associated binding proteins.
Change in costs with the Treatment Inventory of Costs in Psychiatric Patients (Tic-P) | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Change in costs for consumption of health care, costs associated with mental illness and production loss among parents due to psychiatric problems in the child concerning the previous four weeks compared to the four weeks before start of intervention (in Swedish crowns), lower cost is better.

CONTACTS AND LOCATIONS:
Overall Officials: Håkan Jarbin, MD, PhD, Principal Investigator — University Hospital of Lund, Lund University
Locations (1):
- Child and Adolescent Psychiatry, Halmstad, Sweden

IPD SHARING:
Plan to Share IPD: No
The data are shared in an anonymized form within the research group but not beyond the research group.